CLINICAL TRIAL: NCT02540512
Title: Auricular Acupuncture for the Acute Management of Pain in the Emergency Department
Brief Title: Acupuncture for Pain in the Emergency Department
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Traci Marin, Assistant Professor - Research Scientist, Loma Linda University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 15063
Record Dates: First submitted 2015-07-29; First posted 2015-09-04 (Estimated); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Musculoskeletal Pain; Pain
MeSH Terms: conditions — Musculoskeletal Pain; Pain | interventions — Acupuncture, Ear; Acupuncture Therapy; Hydrocodone; Acetaminophen; oxycodone-acetaminophen; Drugs, Generic; Methylcellulose; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Drug Group (Placebo Comparator): Participants randomized into this group will be receiving the standard medical care and "placebo" acupuncture. For the placebo acupuncture procedure, the ASP® needles will be double taped onto the ear in the same anatomical position as the acupuncture groups. The needles will be taped so that the needles will never puncture the skin. The patients will then be given hydrocodone / acetaminophen 5mg/325mg (generic) with a prescription to take home and use as needed.
  Interventions: Device: Acupuncture; Procedure: Placebo Acupuncture; Drug: hydrocodone / acetaminophen 5mg/325mg
- Standard Drug Plus Acupuncture Group (Experimental): The participants in this group will receive auricular acupuncture following the Battlefield Acupuncture Protocol. The patients will then be given hydrocodone / acetaminophen 5mg/325mg (generic) with a prescription to take home and use as needed (in the acupuncture groups, the physician administering the treatment will not know if the patient is receiving the standard drug or the placebo pill). The physician can administer up to 10 needles (5 in each ear) until the patient has a "significant" drop in pain (pain level 0 or 1).
  Interventions: Procedure: Auricular Acupuncture; Device: Acupuncture; Drug: hydrocodone / acetaminophen 5mg/325mg
- Acupuncture Group (Experimental): The participants in this group will receive auricular acupuncture following the Battlefield Acupuncture Protocol. The physician can administer up to 10 needles (5 in each ear) until the patient has a "significant" drop in pain (pain level 0 or 1). The patient will then be given a placebo pill.
  Interventions: Procedure: Auricular Acupuncture; Device: Acupuncture; Drug: Placebo Pill

INTERVENTIONS:
Procedure: Auricular Acupuncture — Aiguille Semi-Permanent (ASP) acupuncture needles will be used following the Battlefield Acupuncture Protocol
  Other Names: Battlefield Acupuncture
  Arms: Acupuncture Group; Standard Drug Plus Acupuncture Group
Device: Acupuncture — ASP Needles: Small, semi-permanent acupuncture needles that will be used for acupuncture in the ear or taped over the ear for placebo.
  Other Names: Aiguille Semi-Permanent (ASP) acupuncture needles
Procedure: Placebo Acupuncture — The ASP needles will be double taped onto the ear for this procedure.
  Arms: Standard Drug Group
Drug: hydrocodone / acetaminophen 5mg/325mg — Narcotic/NSAID medication used as the "standard medical treatment"
  Other Names: Norco (generic)
  Arms: Standard Drug Group; Standard Drug Plus Acupuncture Group
Drug: Placebo Pill — Pills will be filled with methylcellulose and administered as a placebo for this intervention.
  Other Names: methylcellulose (sugar pill)
  Arms: Acupuncture Group

SUMMARY:
The purpose of the study is to test auricular (ear) acupuncture for the acute management of patient pain in the Emergency Department as an alternative and adjunct to standard medical treatment.

Currently, physicians who practice medicine here in the United States only have pharmacological intervention at their disposal as the only available treatment tool they have for the treatment and management of pain, and as a result, painkiller misuse, overdose, and death has become the leading health epidemic in America. American healthcare is in desperate need of alternative and safer ways to prevent prescription painkiller overdoses and to better manage pain. If prescription painkiller dependencies can be avoided at the source, potentially many lives and healthcare dollars can be saved. Acupuncture is an alternative treatment that has been effectively used to treat pain for thousands of years in countries around the world. The National Institutes of Health (NIH) and the United Nations World Health Organization (WHO) have stated that acupuncture is a safe and effective treatment for the management of pain. Supported by many studies illustrating seventy-five to ninety-nine percent effectiveness in treating pain with an instantaneous drop in pain by twenty-five to eighty percent, acupuncture appears to be the safest and most effective option available to manage pain syndromes in the emergency department.

Auricular acupuncture has demonstrated beneficial effects to reduce acute and chronic pain intensity. Specifically, for the thesis of this clinical trial, the investigators hypothesize that auricular acupuncture can be an effective alternative and/or adjunct treatment tool in the civilian emergency department for the acute management of pain.

In order to test the safety and efficacy of using auricular acupuncture in the emergency department, people presenting to the emergency department with pain who are willing to participate in the study will be randomized into three separate groups:

1. Standard medical group (tape on ear + standard medical drug)
2. Standard medical group plus auricular acupuncture (acupuncture + standard medical drug)
3. Auricular acupuncture group (acupuncture + placebo pill)

The design of these groups will allow the investigators to best test the efficacy of auricular acupuncture versus the placebo effect and standard medical care as well as an adjunct to standard medical care. To accomplish the objective of this proposal, the investigators will pursue the following specific aims:

Specific Aim 1: To prove the efficacy of auricular acupuncture over a placebo group in the management of pain syndromes. By having the acupuncture group and sham acupuncture group, the investigators will be able to effectively compare the difference in pain levels with a placebo-group.

Specific Aim 2: To prove that auricular acupuncture is an effective alternative and/or adjunct to standard medical care in the Emergency Department.

By testing the efficacy of acupuncture in conjunction with standard medical treatment, the investigators expect to see a potentiation of analgesic effects, and this will be noted by an increased reduction in pain between the standard medical plus acupuncture group versus the standard group and acupuncture group.

Specific Aim 3: To prove that auricular acupuncture as an effective pain management alternative that decreases short-term prescription painkiller dependency.

Through a series of follow up questionnaires and a medication diary that the investigators will give to the patient prior to discharge, the investigators will track the patient's need and use of additional pain medications post treatment. These surveys will give a good indication as to the effectiveness of auricular acupuncture to reduce a patient's dependency on painkiller drugs in the short-term setting.

DETAILED DESCRIPTION:
All Emergency Department physicians willing to participate in the study will be trained on the Battlefield Acupuncture Protocol through a weekend workshop and training. The acupuncture protocol and training will be taught by consulting expert acupuncturists with extensive training and clinical experience with the protocol. The acupuncturists will be available throughout the duration of the study as consultants for the physicians at any time if they have questions about the treatment and/or protocol.

Patients presenting to the Emergency Department that meet all inclusion and exclusion criteria and are willing to participate in the study, have been screened and triaged appropriately, meet all of the inclusion and exclusion criteria for the study, and have given proper informed consent will be randomized into three separate groups:

1. Standard medical group (tape on ear + standard medical drug)
2. Standard medical group plus auricular acupuncture (acupuncture + standard medical drug)
3. Auricular acupuncture group (acupuncture + placebo pill)

Each group will have the appearance of getting the same treatment, and all participants will be informed prior to treatment of each group they could possibly be in.

This is a single blind study with additional considerations to better limit bias. Prior to treatment, the physician will inform each patient of all of the steps utilized in the procedure. In an attempt to limit bias as much as possible, the physician will not know what treatment group the patient will be placed in until just prior to performing the treatment.

The standard medical drug that will be used for this study is hydrocodone / acetaminophen 5mg/325mg (Norco generic).

This is a single-blind study with extra considerations to limit bias. After informing the patient of the procedure and just prior to performing the treatment, the physician will be presented with a box containing all of the supplies needed for the application of the treatment. Each box will contain the supplies for one of the three groups listed above, and once opening the box, the physician will then perform the appropriate treatment. The physician will not know whether or not the patient will be receiving the standard medical drug or the placebo pill. The physician will only know which type of acupuncture procedure will be performed on the patient.

Richard C. Niemtzow, MD, PhD, MPH is the originator and developer of the Battlefield Acupuncture protocol and technique, and he initiated the use of this protocol with great success in the military. Dr. Niemtzow has also proven great success in treating pain with this protocol in other similar research studies in the past.

The investigational protocol and device that will be tested in this study is The Battlefield Acupuncture Protocol, which uses Gold or Titanium French Aiguille Semi-Permanent (ASP) needles. The French ASP® needles are small, single-use, disposable needles that are designed to stay in the ear for several days and will fall out on their own. The ASP needle is a small needle housed within a small plastic injector that allows the acupuncturist to insert a needle in a rapid manner to decrease discomfort. ASP needles are intended for single use and are manufactured in a sterile environment. After all of the appropriate needles have been placed, the ASP needles will be covered with a small adhesive patch to keep the needles securely in place and to prevent contamination. The needles usually remain in the ear for approximately 4 to 6 days before they fall out on their own.

Following the Battlefield Acupuncture Protocol, patients in the acupuncture group will receive auricular acupuncture by medical acupuncturists using sterile ASP® needles (SEDATELEC; Lyon, France bilaterally in the sequence outlined below:

1. Cingulate Gyrus
2. Thalamus
3. Omega 2
4. Point Zero
5. Shen Men

Appropriate asepsis technique will be used to clean the acupuncture points prior to treatment. After the placement of each needle and before the placement of the next needle, the patient will be instructed to walk thirty feet. If the patient is unable to walk, they will be instructed to move their arms for thirty seconds. If the patient experiences a significant drop in their pain level (down to 0 or 1) after the placement of a needle at a specific point and the subsequent movement, no more needles are inserted. If the patient is still in pain, the procedure is repeated until all of the appropriate acupuncture sites are utilized.

Here is a quick breakdown of the steps for performing the Battlefield Acupuncture Protocol:

1. Assess patient's pain level using the VAS score (0-10).
2. Insert one needle into Point 1 (cingulate gyrus)
3. Instruct patient to walk for 30 seconds. If the patient is unable to walk, instruct them to move their arms for 30 seconds.
4. Reassess patient's pain level. If the patient experiences a significant drop in pain (down to 0 or 1), no more needles will be inserted.
5. If pain does not significantly drop, the next needle will be inserted into the same point in the opposite ear and Step 3 will be repeated.
6. If after the insertion of a needle and completion of Step 3 and the patient does experience a drop in pain but it is not significant (down to 0-1), then the sequence of needles will be continued on that same ear that the patient had the drop in pain until the pain level is down to 0-1. This is called the "dominant ear".

Gold ASP® needles are the preferred needles of choice for the protocol, however, if the patient will be having a MRI performed on them within the next week, titanium ASP® needles will be used instead as they will not interfere with the MRI scan.

The patients will then be instructed to leave the needles and tape on their ear for the next 48 hours, not touch them, and allow the needles to fall out on their own. Prior to leaving the Emergency Department after treatment, the patient will schedule a follow-up appointment 48 hours later that will be conducted at the Loma Linda University Clinical Trial Center where the acupuncture needles will be removed, the last pain assessment will be performed, and the patient will fill out the past trauma history questionnaire.

The patients will be asked a series of short questions regarding their pain level and recent painkiller use and asked to fill out a questionnaire about their past trauma history:

Questionnaires:

Patients pain level (utilizing the VAS pain score on a scale of 0-10) and recent painkiller use will be assessed four times during the study, and prior to leaving, patients will be given a medication diary to track their use of painkillers for the following 48 hours after treatment.

1. Prior to treatment (in person at time of triage)
2. Immediately after treatment (patient will fill out an form and drop it in a box prior to leaving)
3. 24 hours after treatment (by phone call)
4. 48 hours after treatment (by in person interview at Loma Linda University Clinical Trial Center)

Patients will also be asked to fill out a questionnaire regarding their past trauma history (see attached questionnaire).

The data collected from this study is as follows: 1. Demographic information, 2. Pain medication use, 3. Pain level, 4. Number of acupuncture needles used for treatment (acupuncture groups), 5. Past trauma history questionnaire.

1. The patient will fill out a form providing their demographic data during the initial screening.
2. During the initial analysis, the patient will be asked how much pain medication they typically use per day. After treatment, the patient will be given a medication diary for them to record their pain medication use over the next two days. The medication use data from the diary will be collected during an over the phone interview performed by the study collaborators.
3. The pain level scoring system that will be used for this study is the Visual Analog Scale (VAS) pain score on a scale of 1-10. The triage nurse will perform the initial recording at time of triage. The patient will do the second recording immediately after treatment as they will fill out a form and drop it in a box prior to leaving the treatment area. The third and fourth pain recordings will be performed by one of the study collaborators who will contact the patients through a follow up interview over the phone.
4. For the patients in the acupuncture groups, the physician will record the number and location of the acupuncture needles used to illicit a positive response in each patient in the patient's chart.

Data Analysis We will compare baseline characteristics between the four treatment groups using X2 tests for categorical variables and independent t test analyses for continuous variables. We will perform a series of these tests to look for differences between groups on a number of relevant baseline variables, including demographic information, intensity of pain, and number of needles used (for acupuncture groups). If the distribution of the four individual pain scores is fairly normal, we will assess changes in pain levels between baseline and follow-ups using independent t tests. We will run nonparametric Kruskal-Wallis tests as well to see whether consistent results will be reached as with the independent, parametric t test. If the same conclusions are reached with both tests, we will assess all outcome measures of pain administered at baseline, immediately after treatment, 24-hours after treatment, and 48-hours after treatment using the independent t test analysis and the intention-to-treat principle. We will calculate effect sizes by taking the difference between the mean changes in pain in the intervention groups and those in the standard care group and dividing it by the SD of the change score in the total population.

Risks and Benefits This is not the first study that has been conducted testing the use of ASP needles for the treatment and management of pain, and ASP needles are approved for use by the FDA.

The potential minor risks and measures to minimize those risks are as follow:

1. There is a minor risk that patients in the placebo group will not experience any relief of pain. Subjects will be made aware of this potential risk prior to giving informed consent. This risk is minor as all subjects will be hemodynamically stable as a part of the inclusion criteria, they will have the opportunity to withdraw from the study at any time if they wish to do so, the physician or nurse can pull the patient from the study if they deem medically necessary, and the study is only 48 hours in duration so as to not cause long-term pain or suffering on any person in the placebo group.
2. Side effects: The most common serious side effect of acupuncture is needle site pain and infection. Acupuncturists will use proper asepsis technique prior to each treatment, and only sterile needles will be used. In case of infection or pain, patients will have the opportunity to come back to the hospital to have the needles removed and to be treated for the infection.
3. Minor confidentiality risk: All subject data will be kept confidential and will be managed with high security. Only the study collaborators will have access to the patient data, and all data will remain locked in files and shredded once used.

Auricular Acupuncture has the potential to provide safe, fast, and effective treatment for the millions of people suffering from pain worldwide. This study has the potential to prove that auricular acupuncture is an acceptable alternative and/or adjunct treatment tool that healthcare providers can use to ease the suffering of people in pain. This study also has the potential to prove auricular acupuncture as an effective tool to reduce the use and dependency on narcotic pain medications.

There are no benefits that will be utilized in this study. All subjects will give informed consent in order to participate in the study.

The training/consulting acupuncturists will be reimbursed for the exact cost of their training and travel expenses.

ELIGIBILITY:
Inclusion Criteria:

* All hemodynamically stable, adult patients presenting to the Emergency Department (ED) with a chief complaint of pain AND a physician diagnosis of acute, non-critical, musculoskeletal pain.
* Musculoskeletal pain includes pain to any bones, muscles, cartilage, or nerves associated with such.
* Patients will be diagnosed by a physician as non-critical meaning they can be treated and sent home without needing to be admitted to the hospital.
* Blood pressure: 90-180/60-110
* Cardiac rate with no dysrhythmias 50-149
* Ventilatory rate 10-35
* Oxygen saturation >87%
* Alert and able to follow commands and respond appropriately

Exclusion Criteria:

* Patients that are altered and/or present with vital signs outside of the inclusion criteria ranges.
* Those deemed in critical condition by triage nurse and/or ER physician.
* Patients with a history of narcotic drug abuse/dependency.
* Patients who have had Battlefield Acupuncture done in the past.
* Pregnant or nursing women (confirmed by a pregnancy test)
* Allergic to adhesive tape, gold, or other needle components
* Allergic to aspirin, NSAIDs, or narcotics
* Patients at risk for complications from indwelling acupuncture needles, such as patients with bleeding disorders, those who are immunosuppressed, or those with liver disease (Hepatitis C, cirrhosis, etc.)

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-07-27 (Estimated); Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity Measure (VAS score 0-10) | 48 hours
  Measurement of patient's pain level over 48 hours (VAS score 0-10)

SECONDARY OUTCOMES:
Recurrence of Pain (VAS score 0-10) | 48 hours
  Monitoring of patient's pain level over 48 hours (VAS score 0-10)
Medication Usage | 48 hours
  Monitoring of patients medication usage over 48 hours with a medication diary which they will take home and fill out each time they use their medication.
Past Trauma History | 48 hours
  Using Center for Disease Control questionnaires to assess past trauma history

CONTACTS AND LOCATIONS:
Overall Officials: Traci Marin, PhD, Principal Investigator — Assistant Professor-Research Scientist

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Asher GN, Jonas DE, Coeytaux RR, Reilly AC, Loh YL, Motsinger-Reif AA, Winham SJ. Auriculotherapy for pain management: a systematic review and meta-analysis of randomized controlled trials. J Altern Complement Med. 2010 Oct;16(10):1097-108. doi: 10.1089/acm.2009.0451. PMID 20954963
- [Background] Bart-Knauer B, Friedl KE. When will acupuncture become a first-line treatment for acute pain management? Mil Med. 2013 Aug;178(8):827-8. doi: 10.7205/MILMED-D-13-00119. No abstract available. PMID 23929041
- [Background] Bodnar RJ. Endogenous opiates and behavior: 2011. Peptides. 2012 Dec;38(2):463-522. doi: 10.1016/j.peptides.2012.09.027. Epub 2012 Oct 3. PMID 23041439
- [Background] Busch V, Zeman F, Heckel A, Menne F, Ellrich J, Eichhammer P. The effect of transcutaneous vagus nerve stimulation on pain perception--an experimental study. Brain Stimul. 2013 Mar;6(2):202-9. doi: 10.1016/j.brs.2012.04.006. Epub 2012 May 7. PMID 22621941
- [Background] Centers for Disease Control. Prescription Painkiller Overdoses in the U.S. (2012). Prescription Painkiller Overdoses in the U.S.,4.
- [Background] Cheng RS, Pomeranz BH. Electroacupuncture analgesia is mediated by stereospecific opiate receptors and is reversed by antagonists of type I receptors. Life Sci. 1980 Feb 25;26(8):631-8. doi: 10.1016/0024-3205(80)90239-8. No abstract available. PMID 6247596
- [Background] Cho, Son, Han: (MRI Neurophysiological evidence of acupuncture mechanisms. Med Acupuncture. 2002: 14: 16-22.
- [Background] Dincer F, Linde K. Sham interventions in randomized clinical trials of acupuncture--a review. Complement Ther Med. 2003 Dec;11(4):235-42. doi: 10.1016/s0965-2299(03)00124-9. PMID 15022656
- [Background] Faircloth AC, Dubovoy A, Biddle C, Dodd-McCue D, Butterworth JF 4th. CME Article: Perceptions of Acupuncture and Acupressure by Anesthesia Providers: A Quantitative Descriptive Study. Med Acupunct. 2016 Apr 1;28(2):79-86. doi: 10.1089/acu.2015.1161. PMID 27158297
- [Background] Fang JQ, Fang JF, Liang Y, Du JY. Electroacupuncture mediates extracellular signal-regulated kinase 1/2 pathways in the spinal cord of rats with inflammatory pain. BMC Complement Altern Med. 2014 Aug 4;14:285. doi: 10.1186/1472-6882-14-285. PMID 25091495
- [Background] Feng Y, Bai L, Ren Y, Wang H, Liu Z, Zhang W, Tian J. Investigation of the large-scale functional brain networks modulated by acupuncture. Magn Reson Imaging. 2011 Sep;29(7):958-65. doi: 10.1016/j.mri.2011.04.009. Epub 2011 May 25. PMID 21616623
- [Background] Ferraz MB, Quaresma MR, Aquino LR, Atra E, Tugwell P, Goldsmith CH. Reliability of pain scales in the assessment of literate and illiterate patients with rheumatoid arthritis. J Rheumatol. 1990 Aug;17(8):1022-4. PMID 2213777
- [Background] Garcia AM. State laws regulating prescribing of controlled substances: balancing the public health problems of chronic pain and prescription painkiller abuse and overdose. J Law Med Ethics. 2013 Mar;41 Suppl 1:42-5. doi: 10.1111/jlme.12037. PMID 23590739
- [Background] Goertz CM, Niemtzow R, Burns SM, Fritts MJ, Crawford CC, Jonas WB. Auricular acupuncture in the treatment of acute pain syndromes: A pilot study. Mil Med. 2006 Oct;171(10):1010-4. doi: 10.7205/milmed.171.10.1010. PMID 17076456
- [Background] Haker E, Egekvist H, Bjerring P. Effect of sensory stimulation (acupuncture) on sympathetic and parasympathetic activities in healthy subjects. J Auton Nerv Syst. 2000 Feb 14;79(1):52-9. doi: 10.1016/s0165-1838(99)00090-9. PMID 10683506
- [Background] Hommer DH. Chinese scalp acupuncture relieves pain and restores function in complex regional pain syndrome. Mil Med. 2012 Oct;177(10):1231-4. doi: 10.7205/milmed-d-12-00193. PMID 23113454
- [Background] Ip, V. (1999). The use of acupuncture for pain relief in a Chinese hospital clinic. Acupuncture In Medicine, 17(2), 101-109.
- [Background] Kawakita K, Funakoshi M. Suppression of the jaw-opening reflex by conditioning a-delta fiber stimulation and electroacupuncture in the rat. Exp Neurol. 1982 Nov;78(2):461-5. doi: 10.1016/0014-4886(82)90063-2. No abstract available. PMID 7140908
- [Background] King HC, Hickey AH, Connelly C. Auricular acupuncture: a brief introduction for military providers. Mil Med. 2013 Aug;178(8):867-74. doi: 10.7205/MILMED-D-13-00075. PMID 23929047
- [Background] Liu J, Qin W, Guo Q, Sun J, Yuan K, Dong M, Liu P, Zhang Y, von Deneen KM, Liu Y, Tian J. Divergent neural processes specific to the acute and sustained phases of verum and SHAM acupuncture. J Magn Reson Imaging. 2011 Jan;33(1):33-40. doi: 10.1002/jmri.22393. PMID 21182118
- [Background] Mohler, Stanley R. "Acupuncture Helps in Treating Medical Problems." Human Factors & Aviation Medicine. Flight Safety Foundation: September-October 2002, Vol. 49 No. 5
- [Background] Moseley JB, O'Malley K, Petersen NJ, Menke TJ, Brody BA, Kuykendall DH, Hollingsworth JC, Ashton CM, Wray NP. A controlled trial of arthroscopic surgery for osteoarthritis of the knee. N Engl J Med. 2002 Jul 11;347(2):81-8. doi: 10.1056/NEJMoa013259. PMID 12110735
- [Background] Napadow V, Edwards RR, Cahalan CM, Mensing G, Greenbaum S, Valovska A, Li A, Kim J, Maeda Y, Park K, Wasan AD. Evoked pain analgesia in chronic pelvic pain patients using respiratory-gated auricular vagal afferent nerve stimulation. Pain Med. 2012 Jun;13(6):777-89. doi: 10.1111/j.1526-4637.2012.01385.x. Epub 2012 May 8. PMID 22568773
- [Background] NIH Consensus Conference. Acupuncture. JAMA. 1998 Nov 4;280(17):1518-24. PMID 9809733
- [Background] Shepherd J. Combating the prescription painkiller epidemic: a national prescription drug reporting program. Am J Law Med. 2014;40(1):85-112. doi: 10.1177/009885881404000103. PMID 24844043
- [Background] Pickett, H. (2011). Battlefield acupuncture. Journal Of Chinese Medicine, (96), 12-17.
- [Background] Pomeranz B, Chiu D. Naloxone blockade of acupuncture analgesia: endorphin implicated. Life Sci. 1976 Dec 1;19(11):1757-62. doi: 10.1016/0024-3205(76)90084-9. No abstract available. PMID 187888
- [Background] Qu F, Zhou J. Electro-acupuncture in relieving labor pain. Evid Based Complement Alternat Med. 2007 Mar;4(1):125-30. doi: 10.1093/ecam/nel053. Epub 2006 Aug 17. PMID 17342250
- [Background] Roberts, C. (2008). Easing Pain with Acupuncture. Soldiers, 63(7), 36-37.
- [Background] Sator-Katzenschlager SM, Scharbert G, Kozek-Langenecker SA, Szeles JC, Finster G, Schiesser AW, Heinze G, Kress HG. The short- and long-term benefit in chronic low back pain through adjuvant electrical versus manual auricular acupuncture. Anesth Analg. 2004 May;98(5):1359-64, table of contents. doi: 10.1213/01.ane.0000107941.16173.f7. PMID 15105215
- [Background] Spielman, F.J. "Acupuncture: What's the Point?" American Journal of Anesthesiology Volume 28 (2001): 306-308.
- [Background] Substance Abuse and Mental Health Services Administration Public Health Service U.S. Department of Health and Human Services. Summary of the 2009 National Survey on Drug Use and Health. J Pain Palliat Care Pharmacother. 2010 Dec;24(4):434-8. No abstract available. PMID 21438417
- [Background] Volkow ND, McLellan TA, Cotto JH, Karithanom M, Weiss SR. Characteristics of opioid prescriptions in 2009. JAMA. 2011 Apr 6;305(13):1299-301. doi: 10.1001/jama.2011.401. No abstract available. PMID 21467282
- [Background] White P, Lewith G, Hopwood V, Prescott P. The placebo needle, is it a valid and convincing placebo for use in acupuncture trials? A randomised, single-blind, cross-over pilot trial. Pain. 2003 Dec;106(3):401-409. doi: 10.1016/j.pain.2003.08.013. PMID 14659523
- [Background] WHO. The World Health Organization Viewpoint on Acupuncture. <www.sd- acupuncture.com/articles.html>. Aug. 13, 2002.
- [Background] Yoo YC, Oh JH, Kwon TD, Lee YK, Bai SJ. Analgesic mechanism of electroacupuncture in an arthritic pain model of rats: a neurotransmitter study. Yonsei Med J. 2011 Nov;52(6):1016-21. doi: 10.3349/ymj.2011.52.6.1016. PMID 22028168
- [Background] Zhang AL, Parker SJ, Smit de V, Taylor DM, Xue CC. Acupuncture and standard emergency department care for pain and/or nausea and its impact on emergency care delivery: a feasibility study. Acupunct Med. 2014 Jun;32(3):250-6. doi: 10.1136/acupmed-2013-010501. Epub 2014 Mar 7. PMID 24610638
- [Background] Zhang Y, Zhang RX, Zhang M, Shen XY, Li A, Xin J, Ren K, Berman BM, Tan M, Lao L. Electroacupuncture inhibition of hyperalgesia in an inflammatory pain rat model: involvement of distinct spinal serotonin and norepinephrine receptor subtypes. Br J Anaesth. 2012 Aug;109(2):245-52. doi: 10.1093/bja/aes136. Epub 2012 May 23. PMID 22628394